CLINICAL TRIAL: NCT05758701
Title: Dual Energy CT Decreased IV Contrast Dose Imaging for TAVR
Brief Title: CT TAVR Abdomen Study
Acronym: CT TAVR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Vikas Kundra, Chief of Oncologic Imaging, Dept. of Radiology and Nuclear Medicine, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HP-00104800
Record Dates: First submitted 2023-02-13; First posted 2023-03-07 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Transcatheter Aortic Valve Replacement
Keywords: Dual energy CT
MeSH Terms: interventions — Iohexol

STUDY DESIGN:
Intervention Model Description: In a standard polyenergetic CT procedure, 100 ml of iodinated contrast is used. Two cohorts of patients will be assessed, the first being given a 1/3rd reduction (33 ml). If satisfactory, a second cohort with 1/4th the standard dosage (25 ml) will be assessed. If unsatisfactory, the IV contrast dose will be increased to 1/2 (50 ml)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): A cohort will be given a 1/3rd reduced dose of iodinated contrast agent (33 ml).
  Interventions: Combination Product: Iodinated Contrast Agent (Omnipaque); Device: Dual Energy CT
- Cohort 2 (Experimental): If imaging with 1/3 dose is satisfactory, a second cohort with 1/4th the standard dosage (25 ml) will be assessed. If images are not satisfactory, contrast dose will be increased to 50 ml.
  Interventions: Combination Product: Iodinated Contrast Agent (Omnipaque); Device: Dual Energy CT

INTERVENTIONS:
Combination Product: Iodinated Contrast Agent (Omnipaque) — Standard dosage of Omnipaque for CT imaging is 100 ml. Cohort will be given a reduced dosage.
Device: Dual Energy CT — Dual energy CT scanners enable monoenergetic CT image reconstruction which allows for improved iodine image contrast.

SUMMARY:
A standard polyenergetic CT (computed tomography) procedure utilizes 100 ml of iodinated contrast. A recent world-wide shortage of iodine based intravenous contrast has highlighted the need to search for alternative methods or doses. Reducing iodinated IV contrast dose can mitigate IV contrast supply shortages and enable significant cost savings for the radiology practice and hospital system. In addition, decreased IV contrast dose can potentially reduce the rate of acute kidney injury, specifically in patients with decreased renal function. The purpose of the study is to determine whether low IV contrast dose CT with monoenergetic reconstruction can be use for presurgical planning of transcatheter valve replacement (TAVR) procedure.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to receive TAVR abdominal CT

Exclusion Criteria:

* cannot undergo CT scan
* Allergy to intravenous contrast not controlled by steroids or benadryl
* GFR<30

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Quality of Images | 18-24 months
  5-point Likert Scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lai MZ, Duzgunes N, Szoka FC. Effects of replacement of the hydroxyl group of cholesterol and tocopherol on the thermotropic behavior of phospholipid membranes. Biochemistry. 1985 Mar 26;24(7):1646-53. doi: 10.1021/bi00328a012. PMID 3839132
- [Background] Gurm HS, Dixon SR, Smith DE, Share D, Lalonde T, Greenbaum A, Moscucci M; BMC2 (Blue Cross Blue Shield of Michigan Cardiovascular Consortium) Registry. Renal function-based contrast dosing to define safe limits of radiographic contrast media in patients undergoing percutaneous coronary interventions. J Am Coll Cardiol. 2011 Aug 23;58(9):907-14. doi: 10.1016/j.jacc.2011.05.023. PMID 21851878